CLINICAL TRIAL: NCT01659632
Title: Gastric Cancer Screening and Alarm Symptoms in Early Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Myung-gui Choi, Professor, The Catholic University of Korea
Other Study IDs: gastric cancer alarm symptom
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Early Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Most of the early gastric cancer are asymptomatic. Symptoms of advanced gastric cancer are weight loss, abdominal pain, nausea, vomiting, anorexia dysphagia, gastrointestinal bleeding. Gastric cancer found according to warning symptoms such as gastrointestinal bleeding, weight loss usually can not be cured. Therefore, early gastric cancer can not be detected and impossible to treatment if endoscopy is performed according to the warning signs. National gastric cancer screening is conducted in men and women of more than 40 years old. The purpose of screening for gastric cancer is discovering a case of possible cure, so increasing the survival rate. The purpose of this study is review of the feasibility of screening for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* gastric cancer patients in St.mary's hospital

Exclusion Criteria:

* gastric lymphoma, gastric GIST patients in St.mary's hospital

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: gastric cancer patients in St.mary's hospital
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-04; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- St. mary's hospital, Seoul, South Korea